CLINICAL TRIAL: NCT02872506
Title: Comparing the Quality of Life of Terminal Ileitis Patients With Crohn's Disease Treated With Anti-TNF or Surgical Resection
Acronym: CASINO
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: investigator decision
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2015_19; 2016-A00019-42 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2016-08-16; First posted 2016-08-19 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Quality of Life
Keywords: Quality of life; Crohn's disease; Ileocecal resection; Anti TNF
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- medical treatment by Anti TNF (Active Comparator): The medical treatment group will be chosen among patients receiving anti-TNF therapy for the first time
  Interventions: Drug: Anti TNF
- ileocecal resection (Active Comparator): The surgical treatment group are the patients operated on for the first time by means of ileocecal resection laparoscopic or laparotomy
  Interventions: Procedure: ileocecal resection

INTERVENTIONS:
Drug: Anti TNF — Patients are admitted to day hospital with blood test less than 7 days. In the absence of contraindications, hydrocortisone infusion 200 mg will be conducted for 15 minutes followed by anti-TNF treatment infusion over 2 hours for the first three sessions. The following infusions of anti-TNF therapy will be on the same terms without hydrocortisone, every 4 to 8 weeks, in doses of 5-10mg/kg. Adverse effect most frequently reported was URTI. The most serious adverse reactions, were a reactivation of hepatitis B, congestive heart failure, serious infection, serum hypersensitivity reactions, blood diseases, systemic lupus erythematosus / lupus-like syndrome, demyelinating disorders, hepatobiliary metabolism disorders. The QOL will be assessed by IBDQ score at the inclusion visit before the first infusion and at 6 months.
  Arms: medical treatment by Anti TNF
Procedure: ileocecal resection — The operation is performed by laparoscopy or laparotomy. Hospital stay is on average 6 days. Preparation for the intervention is sometimes required 3 weeks to 1 month before the procedure to avoid risk situations.The main risk of the intervention is the anastomotic fistula. This risk of anastomotic leakage mainly concerns malnourished patients operated within the context of abdominal sepsis (abscess). An assessment protocol of post-operative pain, every 3 hours, is now well codified in routine surgery. The QOL will be assessed by the IBDQ score before surgery and at 6 months.
  Arms: ileocecal resection

SUMMARY:
Compare the quality of life at 6 months between 2 populations of patients followed for terminal ileitis of Crohn's disease treated with anti-TNF or ileocecal resection.

DETAILED DESCRIPTION:
Two groups of patients suffering from Crohn's terminal ileitis will be matched by sex, age (A2, A3), the time evolution of the disease, the length of the diseased ileal segment (less than 10 cm; 10 to 30; 30 to 50 cm) and the Montreal classification (B1, B2). The medical treatment group will be chosen among patients receiving anti-TNF therapy for the first time. The surgical group are the patients operated on for the first time by means of ileocecal resection by laparoscopy or laparotomy without any severity criteria or perianal lesions and do not require prophylactic treatment of recurrence.

ELIGIBILITY:
Inclusion Criteria:

* isolated Crohn's ileitis without history of bowel resection and never previously been treated with anti-TNF
* Men and woman over 18 years
* Patient with social security cover
* reapproved indication during multidisciplinary meeting
* Patient able to receive clear information in written and oral
* Informed consent signed by the patient

Exclusion Criteria:

* Prophylactic treatment of recurrence before endoscopic control at the 6th postoperative month.
* Contraindication to Anti-TNF after the initial lap works.
* The side effects of surgery or anti-TNF are not exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09 (Estimated); Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
quality of life (QoL) by Inflammatory Bowel Disease Questionnaire | at 6 months from the beginning of medical treatment or surgical resection
  comparing the quality of life (QoL) by Inflammatory Bowel Disease Questionnaire (IBDQ) at 6 months between 2 populations of patients followed for Crohn's terminal ileitis treated with anti-TNF or operated on by means of ileocecal resection

SECONDARY OUTCOMES:
Inflammatory Bowel Disease Questionnaire (IBDQ) | at baseline (beginning of medical treatment or surgical resection), at 6 months
  Inflammatory Bowel Disease Questionnaire (IBDQ) at 6 months between 2 populations of patient
Crohn's disease activity index (CDAI) | at baseline, at 6 months
Length of small intestine segment resection | at baseline
  Length of small intestine segment <10 cm 10 to 30 cm 30 to 50 cm
Duration of hospital stay | at baseline
Clavien-Dindo classification of surgical complications | at baseline, at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Zerbib, MD, PhD, Principal Investigator — University Hospital, Lille

IPD SHARING:
Plan to Share IPD: No